CLINICAL TRIAL: NCT06877429
Title: Is the Diurnal Variation in Circulating Levels of Cortisol Reflected in Follicular Fluid of Preovulatory Follicles Close to Ovulation?
Status: Not yet recruiting | Type: Observational
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Research Director, ART Fertility Clinics LLC
Other Study IDs: 2502-ABU-005-BL
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: ovarian stimulation; cortisol; cortisone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: will have oocyte retrieval at 8.00 a.m.: Ovarian stimulation for both groups (Group A and B): 150 mcg Corifollitropin-Alpha (Elonva®, MSD) will be started in the afternoon of day 2/3 of the cycle. To inhibit premature LH surge, daily GnRH - antagonist (Orgalutran® 0,25mg, NV Organon) will be administered from the morning of day 6 of stimulation. From day 8 onwards, recFSH (Puregon, NV, The Netherlands) will be started and the dosage will be adjusted to the patients response. Final oocyte maturation will be achieved by administration of a dual trigger (5.000 IU of HCG (Pregnyl®,NV Organon) plus 0.3 mg of GnRH-agonist) as soon as ≥ 3 follicles ≥ 17 mm are present.
  In case that patients are at risk of ovarian hyperstimulation (OHSS), defined as more than 20 follicles above 12 mm, patients will NOT receive hCG but only GnRH-agonist as trigger medication.
  Oocyte retrieval will be carried out 36 hours after HCG administration. Previous studies have described ICSI and IVF procedures in detail (Van Steirteghem et al, 1993; Devroey
  Interventions: Procedure: Time of OPU
- Group B: will have oocyte retrieval at 8.00 p.m.: Ovarian stimulation for both groups (Group A and B): 150 mcg Corifollitropin-Alpha (Elonva®, MSD) will be started in the afternoon of day 2/3 of the cycle. To inhibit premature LH surge, daily GnRH - antagonist (Orgalutran® 0,25mg, NV Organon) will be administered from the morning of day 6 of stimulation. From day 8 onwards, recFSH (Puregon, NV, The Netherlands) will be started and the dosage will be adjusted to the patients response. Final oocyte maturation will be achieved by administration of a dual trigger (5.000 IU of HCG (Pregnyl®,NV Organon) plus 0.3 mg of GnRH-agonist) as soon as ≥ 3 follicles ≥ 17 mm are present.
  In case that patients are at risk of ovarian hyperstimulation (OHSS), defined as more than 20 follicles above 12 mm, patients will NOT receive hCG but only GnRH-agonist as trigger medication.
  Oocyte retrieval will be carried out 36 hours after HCG administration. Previous studies have described ICSI and IVF procedures in detail (Van Steirteghem et al, 1993; Devroey
  Interventions: Procedure: Time of OPU

INTERVENTIONS:
Procedure: Time of OPU — OPU procedure either at 8 am or 8 pm

SUMMARY:
Glucocorticoids and especially cortisol exhibit a pronounced diurnal variation. Levels peak around 8 am and may decrease around two to three times during the day reaching a nadir during the evening and early in the night.

Ovulation has been described as a controlled inflammatory event. Following release of the oocyte, termination of the inflammatory reaction needs to take place in order for the follicle and the developing corpus luteum to avoid further damage. It has been suggested, that locally enhanced cortisol availability may play a role in limiting tissue damage and by acting as anti-inflammatory agents mediating repair and remodeling. The aim of the present study is evaluate the concentration of cortisol and cortisone in sets of serum and follicular fluid samples collected simultaneous and at different times of the day (8.00 a.m. and 8.00 p.m.) and compare the levels with the time of the day at which they are collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for IVF / ICSI - treatment

  * Age ≥ 18 years and ≤ 35 years
  * Body weight: 19 - 29 kg/m2
  * Ovarian reserve parameters in the adequate age - range, determined by Anti-Muellerian-Hormone (AMH) and Antral Follicle Count (AFC) (Shebl 2011, Hamdine 2015)
  * Regular cycle (25-35 days)

Exclusion Criteria:

* Age < 18 years and > 35 years

  * Body weight < 60 kg and > 90 kg
  * Ovarian reserve parameters outside the adequate age - range, determined by Anti-Muellerian-Hormone (AMH) and Antral Follicle Count (AFC) (Shebl 2011, Hamdine 2015)
  * Proven poor responder in preceding IVF-treatment-cycle, according to the Bologna criteria: at least two of the following three features must be present:

    (i) Advanced maternal age (≥40 years) or any other risk factor for POR (poor ovarian response) (ii) A previous POR (≤3 oocytes with a conventional stimulation protocol) (iii) An abnormal ovarian reserve test (i.e. AFC < 5-7 follicles or AMH < 0.5 -1.1 ng/ml)
  * Two episodes of POR after maximal stimulation are sufficient to define a patient as a poor responder in the absence of advanced maternal age or abnormal ORT
  * Diagnosis of polycystic ovarian syndrome (PCOS), according to Rotterdam criteria
  * Endometriosis stage 3 or 4 AFS (American Fertility Society)
  * Irregular cycle (< 25 days and > 35 days)
  * Treatment with GnRH-analogues during the previous 6 months
  * Intake of contraceptive pill (OCP) or any hormonal treatment during the last 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who undergo ovarian stimulation for IVF/ICSI at ART Fertility Clinic Abu Dhabi
Study Population: Healthy women
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the concentration of cortisol and cortisone in serum and follicular fluid samples collected at 8 am versus collection at 8 p.m. | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Evaluate the concentration of sex-steroids and cortisol metabolites in follicular fluid samples collected at 8 am versus collection at 8 p.m. | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ART Fertility Clinics LLC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided
upon request

REFERENCES:
- [Background] Yong PY, Thong KJ, Andrew R, Walker BR, Hillier SG. Development-related increase in cortisol biosynthesis by human granulosa cells. J Clin Endocrinol Metab. 2000 Dec;85(12):4728-33. doi: 10.1210/jcem.85.12.7005. PMID 11134135
- [Background] Tetsuka M, Thomas FJ, Thomas MJ, Anderson RA, Mason JI, Hillier SG. Differential expression of messenger ribonucleic acids encoding 11beta-hydroxysteroid dehydrogenase types 1 and 2 in human granulosa cells. J Clin Endocrinol Metab. 1997 Jun;82(6):2006-9. PMID 9177422
- [Background] Yding Andersen C, Morineau G, Fukuda M, Westergaard LG, Ingerslev HJ, Fiet J, Byskov AG. Assessment of the follicular cortisol:cortisone ratio. Hum Reprod. 1999 Jun;14(6):1562-8. PMID 10357976
- [Background] Shebl O, Ebner T, Sir A, Schreier-Lechner E, Mayer RB, Tews G, Sommergruber M. Age-related distribution of basal serum AMH level in women of reproductive age and a presumably healthy cohort. Fertil Steril. 2011 Feb;95(2):832-4. doi: 10.1016/j.fertnstert.2010.09.012. PMID 20970126
- [Background] Hamdine O, Eijkemans MJ, Lentjes EW, Torrance HL, Macklon NS, Fauser BC, Broekmans FJ. Ovarian response prediction in GnRH antagonist treatment for IVF using anti-Mullerian hormone. Hum Reprod. 2015 Jan;30(1):170-8. doi: 10.1093/humrep/deu266. Epub 2014 Oct 29. PMID 25355590